CLINICAL TRIAL: NCT02145585
Title: Completely Automated Robotic Pharmacological Anesthesia System for Patients Undergoing Elective Cardiac Surgery: a Pilot Study
Brief Title: Robotic Pharmacological Anesthesia System for Elective Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX RNI 01/2014
Record Dates: First submitted 2014-05-14; First posted 2014-05-23 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Robotic pharmacological anesthesia; Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Robotic pharmacological system: Robotic pharmacological system/Automated anesthesia delivery system
  Interventions: Device: Test of pharmacologic anesthesia robot (labVIEW® software)

INTERVENTIONS:
Device: Test of pharmacologic anesthesia robot (labVIEW® software)

SUMMARY:
Closed loop systems for anaesthesia have been shown to be more efficient than manual administration and than Target Control Infusion systems (TCI). So far, there is only one single-center study demonstrating that a system using simultaneously three closed loops for each component of anaesthesia (hypnosis, analgesia and muscle relaxation) is possible, safe and is more efficient than manual administration of anaesthetic drugs. Although the results of this study are very encouraging, they are limited by its sample of patients recruited for non-cardiac surgery only.

The hypothesis of the present trial is that cardiac anesthesia using a completely automated anesthesia delivery system, encompassing each components of anesthesia (hypnosis, analgesia and muscle relaxation) is feasible, safe and reliable.

Thus, the objective of the present trial is to test this pharmacologic anesthesia robot on patients scheduled for elective cardiac surgical procedures with extracorporeal circulation.

Hypnosis is monitored during the surgery according to the brain activity values provided by an objective monitoring parameter, called Bispectral Index (BIS).

A BIS target of 45 is aimed trough the surgery. Performance of propofol hypnosis will be determined clinically by recording the % of sedation time during which the actual BIS is within 10% of the target BIS (excellent control), within 11 -20% (good control), between 21-30% (fair control) and beyond 30% of target (inadequate control).

ELIGIBILITY:
Inclusion Criteria:

* Elective patients
* Patients scheduled to receive an extracorporeal circulation
* Patients aged 18 and older

Exclusion Criteria:

* Minor
* Unable to provide informed consent
* Comatose patients
* Patients with dementia
* Patient who underwent neurosurgery
* Pregnant women
* Patient with muscle disease
* Allergy to Propofol and/or remifentanil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery with extracorporeal circulation
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Performance of closed-loop system for propofol administration defined as the efficacy to maintain Bispectral Index (BIS) as close to the target of 45 as possible. | at inclusion (day 0)
  Hypnosis is monitored during the surgery according to the brain activity values provided by an objective monitoring parameter, called Bispectral Index (BIS).

CONTACTS AND LOCATIONS:
Overall Officials: Cédrick ZAOUTER, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Hôpital Haut Lévêque, Pessac, France